CLINICAL TRIAL: NCT03118479
Title: Effect of Varying Testosterone Levels on Insulin Sensitivity in Men With Idiopathic Hypogonadotropic Hypogonadism
Brief Title: Effect of Varying Testosterone Levels on Insulin Sensitivity in Men With Idiopathic Hypogonadotropic Hypogonadism (IHH)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Because the PI left the institution.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Frances Hayes, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2009 - P - 001874
Record Dates: First submitted 2010-07-14; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Hypogonadotropic Hypogonadism; Kallmann Syndrome
Keywords: IHH; KS; Idiopathic hypogonadotropic hypogonadism; GnRH deficiency
MeSH Terms: conditions — Hypogonadism; Kallmann Syndrome; Idiopathic Hypogonadotropic Hypogonadism | interventions — Anastrozole; Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Androgen only addback (Experimental): Anastrozole 10 mg orally once daily for 3 months Testosterone gel 7.5 g transdermally daily for 3 months.
  Interventions: Drug: Anastrozole Pill; Drug: Testosterone
- Combined sex steroid addback (Experimental): Placebo (sugar pill) tablet once daily for 3 months Testosterone gel 7.5 g transdermally daily for 3 months.
  Interventions: Drug: Testosterone; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Anastrozole Pill — 10 mg of Anastrozole to be taken daily for 3 months.
  Other Names: Arimidex (anastrozole)
  Arms: Androgen only addback
Drug: Testosterone — Androgel 7.5 g to be applied transdermally daily for 3 months.
  Other Names: Androgel
Drug: Placebo Oral Tablet — One tablet to be taken daily for 3 months
  Arms: Combined sex steroid addback

SUMMARY:
The investigators are doing this research study to look at the relationship between testosterone (the main sex hormone in men) and insulin (the hormone that controls blood sugar levels) in men with Idiopathic Hypogonadotropic Hypogonadism (IHH).

The investigators hypothesize that normalizing testosterone levels in men with IHH enhances insulin sensitivity, reduces visceral fat, increases lean body mass, and improves the lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic hypogonadotropic hypogonadism or Kallmann Syndrome
* mean testosterone level less than 300 ng/dl
* stable weight for the previous 3 months (no weight change greater than or equal to 10 lbs)
* normal serum TSH
* normal serum prolactin levels

Exclusion Criteria:

* Type 2 diabetes mellitus
* history of diabetes in parents
* sleep apnea
* bleeding disorder
* seeking fertility
* 2 or more cardiovascular risk factors: smoking, hypertension, diabetes, dyslipidemias, family history of cardiovascular disease before age 60.
* history of previous cardiovascular event: myocardial infarction, unstable angina, cerebro-vascular accident.
* illicit drug use/alcohol use (>4 drinks per day)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2010-09-01 (Actual); Study Completion 2010-09-01 (Actual)

PRIMARY OUTCOMES:
Change in glucose tolerance | Change between baseline and 3 months
  Response to 75 g glucose load
Change in insulin sensitivity | Change between baseline and 3 months
  IV glucose tolerance test

SECONDARY OUTCOMES:
Change in visceral fat | Change between baseline and 3 months
  Assessed by CT of abdomen
Change in resting energy expenditure | Change between baseline and 3 months
  Assessed by metabolic monitor

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Pitteloud, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States